CLINICAL TRIAL: NCT05603767
Title: Effects of Receptive Music Therapy Combined With Virtual Reality on Prevailing Symptoms in Patients With Advanced Cancer
Brief Title: Effects of Receptive Music Therapy Combined With Virtual Reality on Prevalent Symptoms in Patients With Advanced Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Austral University, Argentina (Other)
Responsible Party: Principal Investigator, Maria Julia Cremona, Sponsor-Investigator, Austral University, Argentina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P21-069
Record Dates: First submitted 2022-10-11; First posted 2022-11-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Music Therapy
Keywords: Virtual Reality; Paliative Care; Anxiety; Emotional distress; advanced cancer; prevalent symptoms
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: (RMT+ VR) a) Background settings; b) VR video and music selection; c) Listening experience and VR; and e) Return to alert status (Figure 2).60 patients will be included. All of them are treated by the Palliative Care Unit of the Austral University Hospital. Individuals ≥ 18 years of age with advanced cancer defined from the use of the NECPAL-CCOMS Instrument [20]. They can be hospitalized in the medical clinic service (AUH) or in the Integral Care Unit (ICUA) within the hospital, and must sign the informed consent after being duly explained by the principal investigator. Likewise, they must have (1) a minimum previous ESAS-r of at least 7 points in a symptom, (2) they must be able to adopt a posture of at least 45º in bed and a state of alertness and adequate response, (3) they should not present cognitive impairment (measured by Pfeiffer scale [21] > 2 errors) and (4) have functional hearing (with or without hearing aids or other devices).
Who Masked: Care Provider
Masking Description: Patients who agree to participate will be randomized through the "randomlists" web page to the two study groups. The following day the study collaborators will be in charge of taking the preliminary measurements. Afterwards the patient who has been assigned to RMT + VR will receive the session conducted by the principal investigator The control group will receive no intervention and will continue with their usual care. Between 1-2 hours later, both groups will be visited by the collaborators for subsequent measurements. Which will be recorded again by the collaborators the following 24 hours. In no case will the collaborators know whether the patient received the RMT+ VR intervention or was assigned to the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RMT+ VR (Experimental): The patient selects a video with the Oculus Quest headset and music to be played live.
  Interventions: Other: RMT+ VR
- Control (No Intervention): No intervention

INTERVENTIONS:
Other: RMT+ VR — (RMT+ VR). The responsive music therapy session combined with virtual reality involves four stages: a) Background settings; b) VR video and music selection; c) Listening experience and VR; and e) Return to alert status. The therapist will help the patient to select the video to be used for the experience. Utilizing the application created by the research team, the patient will be provided with four possible scenarios. As for the music, patients are asked to choose music that relaxes them the most. Chosen music can be instrumental music (guitar, electric piano or violin) or sung music with harmonic accompaniment (piano or guitar). In both cases the music will be played live.
  Arms: RMT+ VR

SUMMARY:
The present research seeks to determine whether a single responsive music therapy intervention combined with virtual reality (RMT+VR) reduces prevalent symptoms and improves their overall well-being in hospitalized adult patients with advanced oncologic disease receiving palliative care. This is a prospective study of a randomized clinical trial with a control group. The main variables are pain, exhaustion, drowsiness, nausea, loss of appetite, dyspnea, depression, anxiety, sleep and well-being as well as heart rate.

DETAILED DESCRIPTION:
Music therapy has been shown to be effective in hospitalized patients, reducing the level of stress and anxiety, lowering tension, regulating breathing and relieving pain. However, despite the fact that there are many precedents of this type in palliative care, the quality of the evidence is low. The present research seeks to determine whether a single responsive music therapy intervention combined with virtual reality (RMT+VR) reduces prevalent symptoms and improves their overall well-being in hospitalized adult patients with advanced oncologic disease receiving palliative care. This is a prospective study of a randomized clinical trial with a control group. The main variables are pain, exhaustion, drowsiness, nausea, loss of appetite, dyspnea, depression, anxiety, sleep and well-being as well as heart rate. The duration of the study will be 48 hours. After signing the informed consent, patients will be randomized on the first day receiving RMT+VR, or no intervention at all. The variables will be measured on three occasions, before and after each condition, and 24 hours later.

ELIGIBILITY:
Inclusion Criteria:

* All of them are treated by the Palliative Care Unit of the Austral University Hospital.
* Individuals ≥ 18 years of age with advanced cancer defined from the use of the NECPAL-CCOMS Instrument
* They can be hospitalized in the medical clinic service (AUH) or in the Integral Care Unit (ICUA) within the hospital, and must sign the informed consent after being duly explained by the principal investigator.
* Likewise, they must have a minimum previous ESAS-r of at least 7 points in a symptom,
* they must be able to adopt a posture of at least 45º in bed and a state of alertness and adequate response.

Exclusion Criteria:

* they should not present cognitive impairment (measured by Pfeiffer scale [21] > 2 errors)
* have functional hearing (with or without hearing aids or other devices).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-19 (Actual); Primary Completion 2022-10-11 (Actual); Study Completion 2023-10-11 (Estimated)

PRIMARY OUTCOMES:
change in the guiding symptom | up to 48 hours
  main symptom of the patient among the 9 prevalent symptoms included in the ESAS-r scale(pain, fatigue, nausea, depression, anxiety, drowsiness, appetite, well-being, shortness of breath, and sleep), on a numerical scale from 0 to 10 (10 = worst possible).

SECONDARY OUTCOMES:
change in prevalent symptoms (pain, fatigue, nausea, depression, anxiety, drowsiness, appetite, well-being, shortness of breath, and sleep) | up to 48 hours
  on a numerical scale from 0 to 10 (10 = worst possible) ESAS-r scale
change in Anxiety | up to 48 hours
  The State-Trait Anxiety Inventory is a self-report scale with 20 items to assess state anxiety, on a 4-point Likert scale. It has a score ranging from 0 to 60 points. As for the minimum clinically significant change (MCID) for the STAI, it was set at 10 points. Likewise, a cut-off point of 39 or 40 has been suggested to detect clinically significant symptoms.
change in emotional distress | up to 48 hours
  To measure emotional distress or discomfort, the emotional distress screening questionnaire (DME). The DME gives a total score (0 to 20) formed by the sum of the scores of the answers to the questions referring to the assessment of mood and to the assessment of how the patient is coping with the situation.
change in heart rate | up to 24 hours
  finger oximeter

CONTACTS AND LOCATIONS:
Locations (1):
- Agustina, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No